CLINICAL TRIAL: NCT01980004
Title: Does Potassium Citrate Supplementation Reduce Stone Recurrence in Calcium Phosphate Stone Formers With Risk Factors?
Brief Title: Potassium Citrate Supplementation vs. Dietary Counseling
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: closure due to failure to recruit any patients that met study criteria
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Vanderbilt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13-3010
Record Dates: First submitted 2013-11-01; First posted 2013-11-08 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Kidney Stone
MeSH Terms: conditions — Kidney Calculi | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dietary Education (Experimental): Participants in this treatment arm will undergo dietary counseling for the prevention of kidney stone formation.
  Interventions: Other: Dietary Education
- Potassium Citrate and Dietary Education (Experimental): Participants in this treatment arm will undergo potassium citrate supplementation and dietary counseling for the prevention of kidney stone formation.
  Interventions: Dietary Supplement: Potassium Citrate Supplementation; Other: Dietary Education

INTERVENTIONS:
Dietary Supplement: Potassium Citrate Supplementation — 20 mEq taken twice daily
  Arms: Potassium Citrate and Dietary Education
Other: Dietary Education — Dietary counseling will include both a verbal discussion in the clinic regarding increased fluid intake, a moderate calcium rich diet and lemonade therapy as well as receiving a written handout on these topics.

SUMMARY:
The purpose of this study is to compare the role of potassium citrate supplementation with dietary education versus dietary education alone in the reduction of stone risks and events in patients with predominantly calcium phosphate kidney stones.

DETAILED DESCRIPTION:
The prevalence of kidney stone disease in the United States is increasing. Concurrently, an increase in calcium phosphate stone composition is also being observed. Recurrence of kidney stone disease has been reported as high as 50% at five years. Citrate supplementation is widely considered as one of the primary medical cornerstones to decrease kidney stone recurrence. Urinary citrate is a potent inhibitor of calcium stone formation by binding ionic urinary calcium as well as direct inhibition of calcium oxalate formation. Additionally, increased citrate, an alkali, raises urine pH which alters the solubility of certain stone types including uric acid and cystine stones. Potassium citrate supplementation is the primary proven approach to increasing urinary citrate and is a well-established preventive option in stone disease. However, medication treatment can cause epigastric discomfort, frequent large bowel movements and add to the patient's prescription financial burden. Dietary education including lemonade therapy provides natural dietary sources of citrate and may be an alternative to pharmacologic therapy without the associated gastrointestinal symptoms or costs.

The utility of citrate supplementation has not been previously evaluated prospectively in the calcium phosphate stone former. Calcium phosphate stone formation occurs in a more alkaline urine environment. It has been postulated that citrate supplementation could promote calcium phosphate stone occurrence due to its ability to raise urine pH despite the inhibitory effects of increasing urinary citrate. However, this finding has not been observed in limited retrospective studies. The purpose of this investigation is to prospectively evaluate the benefit of citrate supplementation either through potassium citrate treatment with dietary education vs. dietary education alone to reduce stone recurrence in calcium phosphate stone formers with risk factors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years old, being seen at UNC Chapel Hill or Vanderbilt Urology Clinics
2. Documented stone analysis with ≥ 50% calcium phosphate (hydroxyapatite and/or brushite) composition
3. 24 hour urine citrate (≤ 500) on initial evaluation of at least one 24-hour urine study
4. 24 hour urine pH ≥ 6.0 on initial evaluation of at least one 24-hour urine study

Exclusion Criteria:

1. Documented stone analysis with any calcium carbonate or magnesium ammonium phosphate composition
2. Systemic cause for stone disease (primary hyperparathyroidism, complete distal renal tubular acidosis, systemic acidosis, active urinary tract infection)
3. 24 hour urine calcium/kg (> 4) or 24 hour urine calcium/Cr (>140) on initial evaluation of at least one 24-hour urine study
4. Concurrent medication therapy (potassium citrate, sodium citrate, sodium bicarbonate, diuretic, angiotensin-converting enzyme inhibitor, angiotensin II receptor antagonist, topiramate, acetazolamide)
5. Renal insufficiency (GFR ≤ 60)
6. Elevated serum potassium level (≥ 4.5) or hyperkalemia
7. Low serum bicarbonate level (< 24)
8. High serum calcium level (>10)
9. Pregnancy
10. Inability to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-11; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in 24-hour urine parameters | 4-6 weeks from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Davis J Viprakasit, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- North Carolina Memorial Hospital, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Scales CD Jr, Smith AC, Hanley JM, Saigal CS; Urologic Diseases in America Project. Prevalence of kidney stones in the United States. Eur Urol. 2012 Jul;62(1):160-5. doi: 10.1016/j.eururo.2012.03.052. Epub 2012 Mar 31. PMID 22498635
- [Background] Parks JH, Worcester EM, Coe FL, Evan AP, Lingeman JE. Clinical implications of abundant calcium phosphate in routinely analyzed kidney stones. Kidney Int. 2004 Aug;66(2):777-85. doi: 10.1111/j.1523-1755.2004.00803.x. PMID 15253733
- [Background] Mandel N, Mandel I, Fryjoff K, Rejniak T, Mandel G. Conversion of calcium oxalate to calcium phosphate with recurrent stone episodes. J Urol. 2003 Jun;169(6):2026-9. doi: 10.1097/01.ju.0000065592.55499.4e. PMID 12771710
- [Background] Preminger GM. Renal calculi: pathogenesis, diagnosis, and medical therapy. Semin Nephrol. 1992 Mar;12(2):200-16. PMID 1561497
- [Background] Chow K, Dixon J, Gilpin S, Kavanagh JP, Rao PN. Citrate inhibits growth of residual fragments in an in vitro model of calcium oxalate renal stones. Kidney Int. 2004 May;65(5):1724-30. doi: 10.1111/j.1523-1755.2004.00566.x. PMID 15086911
- [Background] Pattaras JG, Moore RG. Citrate in the management of urolithiasis. J Endourol. 1999 Nov;13(9):687-92. doi: 10.1089/end.1999.13.687. PMID 10608522
- [Background] Robinson MR, Leitao VA, Haleblian GE, Scales CD Jr, Chandrashekar A, Pierre SA, Preminger GM. Impact of long-term potassium citrate therapy on urinary profiles and recurrent stone formation. J Urol. 2009 Mar;181(3):1145-50. doi: 10.1016/j.juro.2008.11.014. Epub 2009 Jan 18. PMID 19152932
- [Background] Penniston KL, Steele TH, Nakada SY. Lemonade therapy increases urinary citrate and urine volumes in patients with recurrent calcium oxalate stone formation. Urology. 2007 Nov;70(5):856-60. doi: 10.1016/j.urology.2007.06.1115. Epub 2007 Oct 24. PMID 17919696